CLINICAL TRIAL: NCT03137784
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled 3-period Complete Cross-over Study to Assess the Bronchodilator Effects and Safety of Glycopyrronium Bromide (NVA237) (25 ug and 50 ug o.d.) in Asthma Patients.
Brief Title: Bronchodilator Effects and Safety of Glycopyrronium Bromide (25 ug and 50 ug o.d.) in Asthma
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CQVM149B2204
Record Dates: First submitted 2017-04-24; First posted 2017-05-03 (Actual); Results first posted 2019-01-16 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Asthma
Keywords: asthma,; NVA237,; glycopyrronium bromide; allergic asthma,; allergy triggered asthma,; reactive asthma,; asthma attack,; difficulty breathing
MeSH Terms: conditions — Asthma; Dyspnea | interventions — Glycopyrrolate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- 1(NVA237 50 ug/NVA237 25 ug/placebo) (Other): Treatment sequence: NVA 237 50 ug, 25 ug and placebo
  Interventions: Drug: NVA237 (glycopyrronium bromide); Drug: Placebo
- 2(NVA237 50 ug/placebo/NVA237 25 ug) (Other): Treatment sequence: NVA 237 50 ug, placebo and 25 ug
  Interventions: Drug: NVA237 (glycopyrronium bromide); Drug: Placebo
- 3 (NVA237 25 ug/NVA237 50 ug/placebo) (Other): Treatment sequence: NVA237 25 ug, 50 ug and placebo
  Interventions: Drug: NVA237 (glycopyrronium bromide); Drug: Placebo
- 4 (NVA237 25 ug/placebo/NVA237 50 ug) (Other): Treatment sequence: NVA 237 25 ug, placebo and 50 ug
  Interventions: Drug: NVA237 (glycopyrronium bromide); Drug: Placebo
- 5 (placebo/NVA237 50 ug/ NVA237 25 ug) (Other): Treatment sequence: Placebo, NVA237 50 ug and 25 ug
  Interventions: Drug: NVA237 (glycopyrronium bromide); Drug: Placebo
- 6 (placebo/ NVA237 25 ug/NVA237 50 ug) (Other): Treatment sequence: placebo, NVA237 25 ug and 50 ug
  Interventions: Drug: NVA237 (glycopyrronium bromide); Drug: Placebo

INTERVENTIONS:
Drug: NVA237 (glycopyrronium bromide) — In each treatment arm, patient will receive NVA237 (glycopyrronium bromide) 25 ug and 50 ug dose
Drug: Placebo — In each treatment arm, patient will receive placebo

SUMMARY:
The purpose of this trial is to characterize the bronchodilator effects and safety of 25 ug and 50 ug o.d. NVA237 (glycopyrronium bromide) doses compared to placebo in asthma patients

DETAILED DESCRIPTION:
This study uses a randomized, double-blind, placebo controlled, 3-period cross-over clinical trial design. During a screening epoch patient eligibility will be assessed. The screening epoch will be followed by a 21-day Run-in epoch during which patients will continue their inhaled corticosteroids use but be withdrawn from LABA-treatment and switched to short-acting bronchodilator-rescue medication. After the Run-in period patients will be randomized to one of the 6 treatment sequences and enter the first 7-day study treatment period. Treatment period one is followed by a 10 to 14 days washout period after which patients begin the second 7-day treatment period which is then followed by a second 10 to 14 days washout period followed by the third 7-day treatment period. At the end of each treatment period spirometry will be performed to assess the primary endpoint in terms of trough FEV1. The study population will consist of approximately 144 patients with asthma who have been treated in a stable regimen of ICS/LABA for at least 4 weeks prior to screening.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adult patients aged >= 18 or =< 65 years
* Patients with a diagnosis of asthma for a period of at least 1 year receiving daily treatment of ICS/LABA in a stable regimen for >= 4 weeks
* Pre-bronchodilator FEV1 of >= 50% and =< 80% of the predicted normal value and an increase in FEV1 of 12% and >= 200 ml during reversibility testing

Key Exclusion Criteria:

* Patients who have had an asthma exacerbation that required either treatment with systemic corticosteroids for at least 3 days, or an emergency room visit, or hospital treatment within 6 weeks prior to screening and patients with a history of life-threatening asthma attacks
* Patients who have had a respiratory tract infection within 4 weeks prior to screening.
* Patients who have smoked or inhaled tobacco products within the past 6 month of screening.
* Patients with a history of chronic lung diseases other than asthma, including (but not limited to) chronic obstructive pulmonary disease, bronchiectasis, sarcoidosis, interstitial lung disease, cystic fibrosis, and tuberculosis (unless tuberculosis is confirmed as no longer active by imaging).
* Patients on Maintenance Immunotherapy (desensitization) for allergies for at least 3 months prior to Run-in who are expected to change therapy throughout the course of the study.
* Patients who during the Run-in period are shown to be intolerable to LABA withdrawal.
* Patients who have discontinued LAMA therapy in the past (e.g. due to intolerance or perceived lack of efficacy).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2017-05-04 (Actual); Primary Completion 2017-12-29 (Actual); Study Completion 2017-12-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (19):
- United States (6):
  - Novartis Investigative Site, North Dartmouth, Massachusetts
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Skillman, New Jersey
  - Novartis Investigative Site, Raleigh, North Carolina
  - Novartis Investigative Site, Medford, Oregon
  - Novartis Investigative Site, El Paso, Texas
- Belgium (3):
  - Novartis Investigative Site, Erpent
  - Novartis Investigative Site, Hasselt
  - Novartis Investigative Site, Mechelen
- Germany (5):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Großhansdorf
  - Novartis Investigative Site, Lübeck
  - Novartis Investigative Site, Wiesbaden
- Japan (2):
  - Novartis Investigative Site, Shinjuku-ku, Tokyo
  - Novartis Investigative Site, Toshima-ku, Tokyo
- Latvia (2):
  - Novartis Investigative Site, Daugavpils, LVA
  - Novartis Investigative Site, Riga
- Novartis Investigative Site, Klaipėda, Lithuania

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 1(NVA237 50 ug/NVA237 25 ug/Placebo) | 2(NVA237 50 ug/Placebo/NVA237 25 ug) | 3 (NVA237 25 ug/NVA237 50 ug/Placebo) | 4 (NVA237 25 ug/Placebo/NVA237 50 ug) | 5 (Placebo/NVA237 50 ug/ NVA237 25 ug) | 6 (Placebo/ NVA237 25 ug/NVA237 50 ug)
Started | 24 | 25 | 25 | 24 | 25 | 25
Completed | 22 | 24 | 25 | 24 | 24 | 25
Not Completed | 2 | 1 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Subject/guardian decision | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Non-compliance with study treatment | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All participants randomized to one of six treatment sequences
Arm/Group | All Participants
Number analyzed (Participants) | 148
Age, Continuous [Mean (Standard Deviation); unit: Years] | 47.3 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75
  Male | 73
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 16
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 12
  White | 120
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Trough FEV1 After One Week of Treatment, Point Estimate
Description: To evaluate the bronchodilator effects of NVA237 (25 ug and 50 ug) compared to placebo in terms of trough FEV1 (mean of 23h 15 min and 23 h 45 min post -dose) following 1 week of treatment in the respective treatment period. Trough FEV1 was assessed by performing spirometry measurements in the clinic for each treatment period. For the primary efficacy variable, trough FEV1 is the mean of two measurements taken at 23h 15 min and 23h 45 min post dose.
Time Frame: Following 1 week of treatment
Population: The Full Analysis Set (FAS) consisted of all patients in the randomized Set (RAN) who received at least one dose of study medication. Following the intent-to-treat principle, patients in the FAS were analyzed according to the treatment they were randomized to in the assigned treatment sequence.
Measure: Least Squares Mean (Standard Error); unit: Liters
Groups:
- NVA237 50 ug: NVA237 50 g capsule
- NVA237 25 ug: NVA237 25 μg capsule
- Placebo: Placebo
Arm/Group | NVA237 50 ug | NVA237 25 ug | Placebo
Number analyzed (Participants) | 147 | 146 | 146
Liters | 2.392 (0.0249) | 2.392 (0.0250) | 2.303 (0.0247)
Statistical Analysis 1: Comparison: NVA237 50 ug vs Placebo; Test type: Other — Treatment difference; p < 0.001, Linear Mixed Model; Linear Mixed Model (LMM) = 0.089, 95% CI 2-sided [0.047 to 0.132]
Statistical Analysis 2: Comparison: NVA237 25 ug vs Placebo; Test type: Other; p < 0.001, Linear Mixed Model; Linear Mixed Model (LMM) = 0.090, 95% CI 2-sided [0.047 to 0.132]

2. Secondary Outcome: FEV1 AUC (5 Min-1 h) After One Week of Treatment
Description: To evaluate the bronchodilator effects of NVA237 (25 ug and 50 ug) compared with placebo in terms of Standardized FEV1 AUC following 1 week of treatment in the respective treatment period. FEV1 was measured with spirometry conducted according to internationally accepted standards. The standardized AUC FEV1 was calculated as the sum of trapezoids divided by the length of time over an entire day (AUC 5min-1h)
Time Frame: Following 1 week of treatment
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | NVA237 50 ug | NVA237 25 ug | Placebo
Number analyzed (Participants) | 147 | 146 | 146
Liters | 2.489 (0.0226) | 2.492 (0.0228) | 2.324 (0.0227)
Statistical Analysis 1: Comparison: NVA237 50 ug vs Placebo; Test type: Other — Treatment difference; p < 0.001, Linear Mixed Model; Linear Mixed Model (LMM) = 0.165, 95% CI 2-sided [0.127 to 0.203]
Statistical Analysis 2: Comparison: NVA237 25 ug vs Placebo; Test type: Other — Treatment difference; p < 0.001, Linear Mixed Model; Linear Mixed Model (LMM) = 0.168, 95% CI 2-sided [0.129 to 0.206]

3. Secondary Outcome: FEV1 AUC (5 Min-4 h) After One Week of Treatment
Description: To evaluate the bronchodilator effects of NVA237 (25 ug and 50 ug) compared with placebo in terms of Standardized FEV1 AUC following 1 week of treatment in the respective treatment period. FEV1 was measured with spirometry conducted according to internationally accepted standards. The standardized AUC FEV1 was calculated as the sum of trapezoids divided by the length of time over an entire day (AUC 5min-4h)
Time Frame: Following 1 week of treatment
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | NVA237 50 ug | NVA237 25 ug | Placebo
Number analyzed (Participants) | 147 | 146 | 146
Liters | 2.522 (0.0223) | 2.525 (0.0224) | 2.346 (0.0223)
Statistical Analysis 1: Comparison: NVA237 50 ug vs Placebo; Test type: Other — Treatment difference; p < 0.001, Linear Mixed Model; Linear Mixed Model (LMM) = 0.176, 95% CI 2-sided [0.141 to 0.212]
Statistical Analysis 2: Comparison: NVA237 25 ug vs Placebo; Test type: Other — Treatment difference; p < 0.001, Linear Mixed Model; Linear Mixed Model (LMM) = 0.179, 95% CI 2-sided [0.144 to 0.215]

4. Secondary Outcome: FEV1 AUC (5 Min - 23 h 45 Min) After One Week of Treatment
Description: To evaluate the bronchodilator effects of NVA237 (25 ug and 50 ug) compared with placebo in terms of Standardized FEV1 AUC following 1 week of treatment in the respective treatment period. FEV1 was measured with spirometry conducted according to internationally accepted standards. The standardized AUC FEV1 was calculated as the sum of trapezoids divided by the length of time over an entire day AUC (5 min - 23 h 45 min)
Time Frame: Following 1 week of treatment
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | NVA237 50 ug | NVA237 25 ug | Placebo
Number analyzed (Participants) | 147 | 146 | 146
Liters | 2.443 (0.0226) | 2.450 (0.0227) | 2.304 (0.0226)
Statistical Analysis 1: Comparison: NVA237 50 ug vs Placebo; Test type: Other — Treatment difference; p < 0.001, Linear Mixed Model; Linear Mixed Model (LMM) = 0.139, 95% CI 2-sided [0.106 to 0.173]
Statistical Analysis 2: Comparison: NVA237 25 ug vs Placebo; Test type: Other — Treatment difference; p < 0.001, Linear Mixed Model; Linear Mixed Model (LMM) = 0.146, 95% CI 2-sided [0.112 to 0.179]

5. Secondary Outcome: Peak FEV1 During 4 Hours Post-dose After 1 Week of Treatment
Description: To evaluate the bronchodilator effects of NVA237 (25 ug and 50 ug) compared with placebo in terms of Peak FEV1 following 1 week of treatment in the respective treatment period. FEV1 was measured with spirometry conducted according to internationally accepted standards. The peak effect following 1 week of treatment was defined as the maximum FEV1 during the first 4 hour on that day.
Time Frame: Following 1 week of treatment
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | NVA237 50 ug | NVA237 25 ug | Placebo
Number analyzed (Participants) | 147 | 146 | 146
Liters | 2.621 (0.0228) | 2.630 (0.0229) | 2.457 (0.0228)
Statistical Analysis 1: Comparison: NVA237 50 ug vs Placebo; Test type: Other — Treatment difference; p < 0.001, Linear Mixed Model; Linear Mixed Model (LMM) = 0.164, 95% CI 2-sided [0.127 to 0.201]
Statistical Analysis 2: Comparison: NVA237 25 ug vs Placebo; Test type: Other — Treatment difference; p < 0.001, Linear Mixed Model; Linear Mixed Model (LMM) = 0.174, 95% CI 2-sided [0.137 to 0.211]

6. Secondary Outcome: Trough Forced Vital Capacity (FVC) After 1 Week of Treatment
Description: To evaluate the bronchodilator effects of NVA237 (25 ug and 50 ug) compared with placebo in terms of FVC following 1 week of treatment in respective treatment period. Trough Forced Vital Capacity (FVC) following 7 Days. FVC is the amount of air which can be forcibly exhaled from the lungs after taking the deepest breath possible. FVC was assessed via spirometry
Time Frame: Following 1 week of treatment
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | NVA237 50 ug | NVA237 25 ug | Placebo
Number analyzed (Participants) | 147 | 146 | 146
Liters | 3.509 (0.0268) | 3.530 (0.0269) | 3.472 (0.0267)
Statistical Analysis 1: Comparison: NVA237 50 ug vs Placebo; Test type: Other — Treatment difference; p = 0.079, Linear Mixed Model; Linear Mixed Model (LMM) = 0.036, 95% CI 2-sided [-0.004 to 0.077]
Statistical Analysis 2: Comparison: NVA237 25 ug vs Placebo; Test type: Other — Treatment difference; p = 0.006, Linear Mixed Model; Linear Mixed Model (LMM) = 0.058, 95% CI 2-sided [0.017 to 0.099]

7. Secondary Outcome: Percent Change From Baseline in FEV1/FVC Ratio
Description: To evaluate the bronchodilator effects of NVA237 (25 ug and 50 ug) compared with placebo in terms of FEV1/FVC ratio following 1 week of treatment in respective treatment period
Time Frame: Following 1 week of treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | NVA237 50 ug | NVA237 25 ug | Placebo
Number analyzed (Participants) | 147 | 146 | 146
Percent change | 0.018 (0.0421) | 0.016 (0.0438) | 0.003 (0.0398)

8. Secondary Outcome: Mean Morning Peak Expiratory Flow (PEF) Following the 1-week Treatment Period
Description: A Peak Expiratory Flow (PEF) meter was distributed to patients at Visit 1, to be used to measure PEF twice-daily as directed. During the Screening and Treatment Periods, PEF was measured in the morning and evening every day. the morning PEF was performed within 15 minutes after waking, and the evening PEF approximately 12 hours later. Patients were encouraged to perform morning and evening PEF measurements before the use of any LABA or rescue medication. The highest of 3 values was recorded as the daily personal best. The personal best was used to calculate the mean morning PEF and mean evening PEF value
Time Frame: Following 1 week of treatment
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: L/min
Arm/Group | NVA237 50 ug | NVA237 25 ug | Placebo
Number analyzed (Participants) | 147 | 146 | 146
L/min | 395.09 (2.948) | 393.87 (2.962) | 369.58 (2.958)
Statistical Analysis 1: Comparison: NVA237 50 ug vs Placebo; Test type: Other — Treatment difference; p < 0.001, Linear Mixed Model; Linear Mixed Model (LMM) = 25.51, 95% CI 2-sided [19.22 to 31.79] — LS Mean of change from baseline in mean morning PEF is calculated with the ANCOVA model using treatment, stratification group, dosing schedule, gender, center grouping, smoking status, and baseline mean morning PEF as covariates
Statistical Analysis 2: Comparison: NVA237 25 ug vs Placebo; Test type: Other — Treatment difference; p < 0.001, Linear Mixed Model; Linear Mixed Model (LMM) = 24.29, 95% CI 2-sided [17.99 to 30.59]

9. Secondary Outcome: Mean Evening Peak Expiratory Flow Rate (PEF) Following 1-week Treatment
Description: A Peak Expiratory Flow (PEF) meter was distributed to patients at Visit 1, to be used to measure PEF twice-daily as directed. During the Screening and Treatment Periods, PEF was measured in the morning and evening every day. the morning PEF was performed within 15 minutes after waking, and the evening PEF approximately 12 hours later. Patients were encouraged to perform morning and evening PEF measurements before the use of any LABA or rescue medication. The highest of 3 values was recorded as the daily personal best. The personal best was used to calculate the mean morning PEF and mean evening PEF value collected between assessment Visits. LS Mean of change from baseline in mean morning PEF is calculated with the ANCOVA model using treatment, stratification group, dosing schedule, gender, center grouping, smoking status, and baseline mean morning PEF as covariates
Time Frame: Following 1 week of treatment
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: L/min
Arm/Group | NVA237 50 ug | NVA237 25 ug | Placebo
Number analyzed (Participants) | 147 | 146 | 146
L/min | 409.66 (2.928) | 408.08 (2.934) | 378.72 (2.949)
Statistical Analysis 1: Comparison: NVA237 50 ug vs Placebo; Test type: Other — Treatment difference; p < 0.001, Linear Mixed Model; Linear Mixed Model (LMM) = 30.95, 95% CI 2-sided [25.07 to 36.82] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 2: Comparison: NVA237 25 ug vs Placebo; Test type: Other — Treatment difference; p < 0.001, Linear Mixed Model; Linear Mixed Model (LMM) = 29.37, 95% CI 2-sided [23.47 to 35.26] — [estimate comment as in outcome 8, analysis 1]

10. Secondary Outcome: Mean Daily Number of Puffs of Rescue Medication During 1 Week of Treatment
Description: A day with no rescue medication use is defined from the diary data as any day where the patient recorded no rescue medicine use during the previous 12 hours. daytime and nighttime (combined) number of puffs is defined as the average of the respective number of puffs.
Time Frame: Following 1 week of treatment
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Puffs/day
Arm/Group | NVA237 50 ug | NVA237 25 ug | Placebo
Number analyzed (Participants) | 147 | 146 | 146
Puffs/day | 0.98 (0.094) | 1.02 (0.094) | 1.13 (0.094)
Statistical Analysis 1: Comparison: NVA237 50 ug vs Placebo; Test type: Other — Treatment difference; p = 0.053, Linear Mixed Model; Linear Mixed Model (LMM) = -0.15, 95% CI 2-sided [-0.31 to 0.00]
Statistical Analysis 2: Comparison: NVA237 25 ug vs Placebo; Test type: Other — Treatment difference; p = 0.163, Linear Mixed Model; Linear Mixed Model (LMM) = -0.11, 95% CI 2-sided [-0.27 to 0.05]

ADVERSE EVENTS:
Time Frame: Following 1 week of treatment
Description: AE additional description
Groups:
- NVA237 50 ug: NVA237 50 ug capsule
- NVA237 25 ug: NVA237 25 ug capsule
Arm/Group | NVA237 50 ug | NVA237 25 ug | Placebo
All-Cause Mortality (participants affected / at risk) | 0/147 | 1/146 | 0/146
Serious Adverse Events (participants affected / at risk) | 1/147 | 1/146 | 0/146
Other Adverse Events (participants affected / at risk) | 10/147 | 11/146 | 11/146
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NVA237 50 ug (N=147) | NVA237 25 ug (N=146) | Placebo (N=146)
Patellofemoral pain syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Completed suicide (Psychiatric disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NVA237 50 ug (N=147) | NVA237 25 ug (N=146) | Placebo (N=146)
Nasopharyngitis (Infections and infestations) | 2 | 1 | 3
Upper respiratory tract infection (Infections and infestations) | 1 | 3 | 1
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 2
Dizziness (Nervous system disorders) | 1 | 0 | 2
Headache (Nervous system disorders) | 5 | 2 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-02-07): https://cdn.clinicaltrials.gov/large-docs/84/NCT03137784/SAP_000.pdf
  • Study Protocol (2016-11-01): https://cdn.clinicaltrials.gov/large-docs/84/NCT03137784/Prot_001.pdf